CLINICAL TRIAL: NCT01389310
Title: Post-marketing Safety Surveillance Program in HIV-infected Children Exposed to Atazanavir in Europe
Brief Title: Post-marketing Safety Surveillance Program in Human Immunodeficiency Virus (HIV)-Infected Children Exposed to Atazanavir in Europe
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: PENTA Foundation (Network)
Responsible Party: Sponsor
Other Study IDs: AI424-450
Record Dates: First submitted 2011-07-06; First posted 2011-07-08 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: HIV Infection
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HIV-infected children <18 yrs old - exposed to Atazanavir

SUMMARY:
The purpose of this study is to monitor adverse events in HIV-infected children <18 years old who are exposed to Atazanavir in a real-world setting in Europe.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected children participating in individual prospective paediatric HIV cohorts
* Receive Atazanavir treatment during 01JAN2011 to 30DEC2013
* Age <18 years old on the date starting an Atazanavir-containing regimen
* Have a minimum of 3 months of follow-up

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 249 (Actual)
Dates: Start 2011-07; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Number of Adverse events reported during Atazanavir drug exposure | 36 months
  Timeframe of the study

SECONDARY OUTCOMES:
Pattern of use of Atazanavir | 12-months
  Atazanavir dosage administered, treatment duration (date started, date stopped), reason for dosage adjustment, withdrawal and reason for withdrawal, Ritonavir dose, other antiretroviral drug use, and other concomitant medications
Pattern of use of Atazanavir | 24-months
  Atazanavir dosage administered, treatment duration (date started, date stopped), reason for dosage adjustment, withdrawal and reason for withdrawal, Ritonavir dose, other antiretroviral drug use, and other concomitant medications
Pattern of use of Atazanavir | 36-months
  Atazanavir dosage administered, treatment duration (date started, date stopped), reason for dosage adjustment, withdrawal and reason for withdrawal, Ritonavir dose, other antiretroviral drug use, and other concomitant medications

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (9):
- Hospital St Pierre, Brussels, Belgium
- German Competence Network, Frankfurt, Germany
- Italian Register for HIV-infection in Children, Florence, Italy
- Victor Babes Hospital, Bucharest, Romania
- Spain (2):
  - Spanish Perinatal Cohort, Barcelona
  - Madrid Paediatric HIV Cohort, Madrid
- Swiss Mother and Child HIV Cohort, Basel, Switzerland
- United Kingdom (2):
  - Collaborative HIV Paediatric Study, London
  - European Collaborative Study, London

REFERENCES:
- See also: BMS Clinical Trials Disclosure — http://www.bms.com/clinical_trials/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx
- See also: For FDA Safety Alerts and Recalls refer to the following link: http://www.fda.gov/MEDWATCH/safety.htm — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm